CLINICAL TRIAL: NCT05790837
Title: Workplace Intervention to Reduce Sitting Time, Decrease Musculoskeletal Symptoms, and Improve Cardiometabolic Markers in Sedentary Office Workers: a Randomized Clinical Trial.
Brief Title: Workplace Intervention to Reduce Sitting Time: a Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Superintendencia de Seguridad Social - Gobierno de Chile (Unknown)
Responsible Party: Principal Investigator, Jaime Leppe Zamora, PhD(C) in Epidemiology, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 280-2022
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Sedentary Behavior; Office Workers
Keywords: Sedentary Behavior; Sitting time; Physical activity; Musculoskeletal symptoms; Cardiometabolic biomarkers
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized parallel-group trial. The groups will be recruited from higher education institutions. The length of this study will be six months. Measurements shall be made for both groups at baseline, 3rd, and 6th months.
  The intervention group will receive the computer prompt "Stand up for your Health®" and information about sedentary behaviour. The computer prompt appears when the workers accumulate one hour the work front to screen. The break is two minutes, and one video with exercises starts with instructions for workers during this time.
  The control group will receive only information through the leaflet.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer prompt + Education (CP+E) (Experimental): The intervention group consists of the implementation of the desktop application "Stand up for your Health®" following the model proposed by the Guide to Physical Activity at Work plus education through an information leaflet
  Interventions: Behavioral: Computer prompt "Stand up for your Health®"
- Only Education (OE) (No Intervention): The control group will receive only education through an information leaflet also following the guidelines of the Work Physical Activity Guide on indications to control the time sitting at work.

INTERVENTIONS:
Behavioral: Computer prompt "Stand up for your Health®" — The intervention group consists on the implementation of a desktop application "Stand up for your Health®" computer prompt following the model proposed by the Guide to Physical Activity at Work (34). This app works by showing reminders and asking users to pause their work activity and take an active break. Pauses can be customized and programmed according to the user's preference, allowing control of the time of each pause, between pauses, and the possibility of delaying or interrupting the pause. In this study, the "Stand up for your Health®" app will be scheduled to appear every 60 minutes on the workers' computers and each break will last for 2 minutes. During this resting period, the worker will see a notice or reminder on their screen with a countdown clock. The application allows you to postpone or interrupt directions.
  Arms: Computer prompt + Education (CP+E)

SUMMARY:
The goal of this randomized clinical trial is to determine the effect of the computer prompt to break sitting time in office workers.

The main question is: What is the effect of the computer prompt "Stand Up for Your Health®" plus education on sitting time, musculoskeletal symptoms, cardiometabolic markers, and physical activity in office workers compared with only education? In addition, to determine the level of adherence to the intervention program by identifying barriers and facilitators referred by the participants.

The participants will be divided into two groups, the experimental and the control group. The participants in the experimental group will use the computer prompt on their desktop and receive information about sedentary behaviour, and the control group will receive only information. All participants will wear accelerometers for one week. The musculoskeletal symptoms and cardiometabolic markers will be measured at baseline, 3rd and 6th month.

DETAILED DESCRIPTION:
Sedentary behaviour and physical inactivity are risk factors for noncommunicable diseases related to the work environment. The accumulation of sitting time during the workday is related to musculoskeletal symptoms and worse cardiometabolic indicators.

The purpose of this study is to determine the effect of the "Stand up for your Health®" computer app on sitting time, musculoskeletal symptoms, cardiometabolic markers, and physical activity in office workers. Also, to determine the adherence to the intervention program by identifying barriers and facilitators referred by the participants.

In this 2-arm randomized controlled trial, both groups will be recruited from educational establishments and will be measured at baseline, 3rd, and 6th months. The experimental group will be implementing the "Stand Up for Your Health®" computer app plus educational information, while the control group will only receive educational information.

The same measurements will be completed in both groups during a 6 months follow-up period: sedentary behaviour using the Actigraph accelerometers and the Occupational Sitting and Physical Activity Questionnaire (OSPAQ); musculoskeletal symptoms will be assessed by a pressure pain algometer and the Standardized Nordic Questionnaire of Perception of musculoskeletal Symptoms; and cardiometabolic markers and anthropometric measurements will also be assessed according to protocol.

ELIGIBILITY:
Inclusion Criteria:

* office workers over 18 years of age,
* Full-time employees (≥35 hours per week);
* Spend most of their workday sitting (> 60%). This will be initially self-reported and used as selection criteria prior to the initial consent and measurement visit. This will be later confirmed using accelerometers;
* Work in the same office place during the week; and
* Able to walk without using an assistive device or requiring the assistance of another person.

Exclusion Criteria:

* Pregnant women;
* Desktop workers using a height-adjustable workstation; and
* Office workers sufficiently active according to WHO criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-09-16 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Sedentary behaviour (occupational sitting time) at baseline | During 1 week at T0 (baseline)
  Sedentary behaviour will be objectively assessed using accelerometers Actigraph GT3X per a period of one week. Data will be downloaded and analyzed with ActiLife software.
  Occupational sitting time shall be measured subjectively using the Occupational Sitting and Physical Activity Questionnaire (OSPAQ).
Sedentary behaviour (occupational sitting time) at 3rd month | During 1 week at T1 (3rd month)
  Sedentary behaviour will be objectively assessed using accelerometers Actigraph GT3X per a period of one week. Data will be downloaded and analyzed with ActiLife software.
  Occupational sitting time shall be measured subjectively using the Occupational Sitting and Physical Activity Questionnaire (OSPAQ).
Sedentary behaviour (occupational sitting time) at 6th month | During 1 week at T2 (6th month)
  Sedentary behaviour will be objectively assessed using accelerometers Actigraph GT3X per a period of one week. Data will be downloaded and analyzed with ActiLife software.
  Occupational sitting time shall be measured subjectively using the Occupational Sitting and Physical Activity Questionnaire (OSPAQ).

SECONDARY OUTCOMES:
Cardiometabolic biomarkers - Fasting blood glucose | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Cardiometabolic health outcomes will be carried out following the standardized protocol in this study population. Measurements of fasting blood glucose in milligrams per deciliter (mg/dL) will be collected in blood samples on an empty stomach in the workplace by a trained and certified health professional.
Cardiometabolic biomarkers - Fasting insulin | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Cardiometabolic health outcomes will be carried out following the standardized protocol in this study population. Measurements of fasting insulin in milligrams per deciliter (mg/dL) will be collected in blood samples on an empty stomach in the workplace by a trained and certified health professional.
Cardiometabolic biomarkers - Cortisol | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Cardiometabolic health outcomes will be carried out following the standardized protocol in this study population. Measurements of cortisol in micrograms per deciliter (mcg/dL)will be collected in blood samples on an empty stomach in the workplace by a trained and certified health professional.
Cardiometabolic biomarkers - Triglycerides | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Cardiometabolic health outcomes will be carried out following the standardized protocol in this study population. Measurements of triglycerides in milligrams per deciliter (mg/dL) will be collected in blood samples on an empty stomach in the workplace by a trained and certified health professional.
Cardiometabolic biomarkers - Total cholesterol | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Cardiometabolic health outcomes will be carried out following the standardized protocol in this study population. Measurements of total cholesterol in milligrams per deciliter (mg/dL) will be collected in blood sample on an empty stomach in the workplace by a trained and certified health professional.
Cardiometabolic biomarkers - Low density lipoprotein cholesterol | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Cardiometabolic health outcomes will be carried out following the standardized protocol in this study population. Measurements of low-density lipoprotein (LDL) cholesterol will be collected in a blood sample on an empty stomach in the workplace by a trained and certified health professional.
Cardiometabolic biomarkers - High density lipoprotein cholesterol | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Cardiometabolic health outcomes will be carried out following the standardized protocol in this study population. Measurements of high-density lipoprotein (HDL) cholesterol will be collected in a blood sample on an empty stomach in the workplace by a trained and certified health professional.
  Anthropometric measurements and blood pressure will be assessed in all participants.
Anthropometric measurements - Height | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Anthropometric measurements outcomes will be carried out following the standardized protocol in this study population. Height in meters (m) will be measured using an altimeter.
Anthropometric measurements - Weight | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Anthropometric measurements outcomes will be carried out following the standardized protocol in this study population. Weight in kilograms (kg) will be measured using a digital scale.
Anthropometric measurements - Waist Circumference | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Anthropometric measurements outcomes will be carried out following the standardized protocol in this study population. Waist Circumference in centimeters (cm) will be measured using a tape measure.
Anthropometric measurements - Body Mass Index | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  Anthropometric measurements outcomes will be carried out following the standardized protocol in this study population. Body Mass Index (BMI) in kilograms per square meters (kg/m2) will be calculated using the weight and height outcome measures.
Musculoskeletal symptoms - Pain | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  A pressure pain threshold algometer shall be used as an objective measurement and will provide a quantitative measurement of sensory perception of mechanical stimuli in kilopascal (kPa) units.
Musculoskeletal symptoms - Symptoms | At T0 (baseline), T1 (3rd month) and T2 (6th month)
  The standardized Nordic Questionnaire of perception of musculoskeletal symptoms will be used as a subjective measurement, providing a numerical pain scale.
  All measurements will be performed by a physiotherapist and following a standardized measurement procedure for office workers

CONTACTS AND LOCATIONS:
Overall Officials: Jaime E Leppe Zamora, PhD©, Principal Investigator — Universidad del Desarrollo, Santiago, Region Metropolitana, Chile
Locations (1):
- Universidad Autónoma de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hadgraft NT, Winkler E, Climie RE, Grace MS, Romero L, Owen N, Dunstan D, Healy G, Dempsey PC. Effects of sedentary behaviour interventions on biomarkers of cardiometabolic risk in adults: systematic review with meta-analyses. Br J Sports Med. 2021 Feb;55(3):144-154. doi: 10.1136/bjsports-2019-101154. Epub 2020 Apr 8. PMID 32269058
- [Background] Taylor WC, Williams JR, Harris LE, Shegog R. Computer Prompt Software to Reduce Sedentary Behavior and Promote Physical Activity Among Desk-Based Workers: A Systematic Review. Hum Factors. 2023 Aug;65(5):891-908. doi: 10.1177/00187208211034271. Epub 2021 Aug 15. PMID 34392738
- [Background] Fernandez-Verdejo R, Suarez-Reyes M. [Physical inactivity versus sedentariness: analysis of the chilean national health survey 2016-2017]. Rev Med Chil. 2021 Jan;149(1):103-109. doi: 10.4067/S0034-98872021000100103. Spanish. PMID 34106141
- [Background] Ekelund U, Brown WJ, Steene-Johannessen J, Fagerland MW, Owen N, Powell KE, Bauman AE, Lee IM. Do the associations of sedentary behaviour with cardiovascular disease mortality and cancer mortality differ by physical activity level? A systematic review and harmonised meta-analysis of data from 850 060 participants. Br J Sports Med. 2019 Jul;53(14):886-894. doi: 10.1136/bjsports-2017-098963. Epub 2018 Jul 10. PMID 29991570
- [Background] Ekelund U, Tarp J, Steene-Johannessen J, Hansen BH, Jefferis B, Fagerland MW, Whincup P, Diaz KM, Hooker SP, Chernofsky A, Larson MG, Spartano N, Vasan RS, Dohrn IM, Hagstromer M, Edwardson C, Yates T, Shiroma E, Anderssen SA, Lee IM. Dose-response associations between accelerometry measured physical activity and sedentary time and all cause mortality: systematic review and harmonised meta-analysis. BMJ. 2019 Aug 21;366:l4570. doi: 10.1136/bmj.l4570. PMID 31434697
- [Background] Parry SP, Coenen P, Shrestha N, O'Sullivan PB, Maher CG, Straker LM. Workplace interventions for increasing standing or walking for decreasing musculoskeletal symptoms in sedentary workers. Cochrane Database Syst Rev. 2019 Nov 17;2019(11):CD012487. doi: 10.1002/14651858.CD012487.pub2. PMID 31742666
- [Background] Nunes AMP, Moita JPAM, Espanha MMMR, Petersen KK, Arendt-Nielsen L. Pressure pain thresholds in office workers with chronic neck pain: A systematic review and meta-analysis. Pain Pract. 2021 Sep;21(7):799-814. doi: 10.1111/papr.13014. Epub 2021 May 6. PMID 33829681
- [Background] Waongenngarm P, Areerak K, Janwantanakul P. The effects of breaks on low back pain, discomfort, and work productivity in office workers: A systematic review of randomized and non-randomized controlled trials. Appl Ergon. 2018 Apr;68:230-239. doi: 10.1016/j.apergo.2017.12.003. Epub 2017 Dec 8. PMID 29409639